CLINICAL TRIAL: NCT04080713
Title: An Open-label Study Investigating the Pharmacokinetic Profile and Safety of Single Oral Dose of Budesonide Prolonged Release Tablets 9mg (Cortiment® MMX) in Healthy Indian Subjects Under Fasting Condition
Brief Title: Cortiment® MMX Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 000326
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Healthy
Keywords: Budesonide; Healthy; Pharmacokinetic
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Budesonide (Experimental)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Budesonide 9 mg prolonged release tablet
  Other Names: Cortiment® MMX

SUMMARY:
Budesonide is a well-known and well-characterised locally acting glucocorticosteroid with comparable efficacy to that of conventional glucocorticosteroids, but with fewer systemic side effects due to its low bioavailability following oral administration.

There are no benefits for subjects participating in this pharmacokinetic (PK) profile and safety study. This is an open-label study to investigate the PK profile and safety of single oral dose of budesonide prolonged release tablets (9 mg, Cortiment® MMX [multi-matrix system]) in healthy subjects in Indian population.

Two study visits are planned: One out-patient visit (screening) and one residential session consisting of three consecutive nights (admission to the clinical investigation unit at least 12 hours before dosing and discharge approximately 60 hours after dosing). End-of-study assessments will be performed before discharge from the clinical investigation unit in the single dosing period. Subjects should be in the fasted state for at least 10 hours pre-dose.

Number of subjects planned in total in the study are 24 men and women, with a minimum requirement of 7 women. The safety assessments comprise of adverse events (AEs), vital signs, electrocardiogram (ECG) and clinical laboratory variables. Adverse events will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Indian men and women between18-45 (both inclusive) years of age (at the time of signed/ thumb impression informed consent).
* Body mass index (BMI) between 18.5 kg/m^2 and 29.9 kg/m^2 (both inclusive) and body weight between 50 kg and 100 kg.
* Negative hepatitis screen including hepatitis B surface antigen (HBsAg) and/or hepatitis C virus (HCV) antibodies at screening.
* Negative test result for human immunodeficiency virus (HIV) (I and II) antibody.
* Healthy according to medical history (including surgical history), physical examination, 12-lead ECG, chest X-ray recordings (postero-anterior view), vital sign (sitting blood pressure, pulse rate and body temperature), and laboratory profile of blood and urine at screening.
* Negative serum pregnancy test (for females) at screening and on Day -1.
* Regular intestinal function; no constipation and no diarrhea.
* Has given written informed consent prior to any study-related activity is performed.
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study.
* Negative alcohol test, urine drug screen test on the day of screening and the day before dosing.
* Non-smokers.
* Agree to use double-barrier contraception or intra-uterine device, intra-uterine system, combined oral contraceptive pill associated with inhibition of ovulation (oral, intravaginal, transdermal), progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) during the study if not abstinent. Previous surgical sterilization of subject or their sexual partner (bilateral tubal ligation, vasectomy) also represents a permissible form of contraception. Methods of double barrier contraception include use of the male condom together with female condom or cervical cap or diaphragm.

Exclusion Criteria:

* Allergy: Ascertained or presumptive hypersensitivity to the active principle, lecithin (derived from soya oil, peanut oil) and/or other formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study.
* Diseases: Presence or relevant history of renal, hepatic, gastrointestinal (GI), cardiovascular, haematological, respiratory or any other body system, any recent or ongoing infections or endocrine or neurologic diseases that may interfere with the aim of the study. Particularly, history of GI diseases, inflammatory bowel disease (IBD), intolerance to lactose; neoplasias.
* Medications: medication, including over-the-counter (OTC) and CYP3A4 inducers/inhibitors or herbal medication, during 2 weeks or five half-lives of the drug, whichever is longer, prior to screening; in particular, drugs affecting GI physiology. Allowed medications included acetaminophen/paracetamol and cromoglycate eye drops according to label, hormonal contraceptives for fertile women.
* Previous or current budesonide treatment.
* Use of live vaccine within 4 weeks prior to dosing.
* Life style: history (within the last two years) or present abuse of drug, alcohol [defined as regular intake of more than 14 units weekly for men /7 units weekly for women - one unit of alcohol equals about 300 mL of beer or lager, one glass (100 mL) of wine, or 25 mL spirits].
* Current smokers or subjects who have smoked within last six months prior to start of the study.
* Consumption of Grapefruits or its products within a period of one-week prior to receiving the study drug.
* Consumption of poppy seeds (e.g., poppy cake) and betel nuts at least seven days at least seven days before receiving the trial drug.
* A high daily consumption of caffeine-containing beverages (e.g., more than five cups of coffee or equivalent) with a risk of withdrawal. symptoms arising during the study that may have confounded the safety evaluation.
* Female subjects who are pregnant, breastfeeding or intend to become pregnant.
* Any medical or surgical condition that may interfere with the absorption, distribution, metabolism, or excretion of the drug, as judged by the investigator.
* Acute illness within two weeks prior to screening.
* Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.
* Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication.

If investigational medicinal product is received within 90 days where there is no blood loss except safety lab testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.

* A mental condition, the lack of decision-making ability, dementia or a speech handicap, which, in the judgement of the Investigator, would impair the participation of the subjects in the study.
* Any other reasons, which will make clinical study participation inappropriate with the decision of the investigator.
* The presence of clinically significant abnormal laboratory values during screening.
* Difficulty in swallowing solids dosage forms like tablets or capsules.
* Previous participation in a budesonide study.
* History of diabetes and/or hyperglycemia.
* History of menstrual disturbances (for females).
* History of hypercorticism.
* History of ophthalmological disorders (e.g. glaucoma).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum plasma concentration observed (Cmax) | Up to 60 hours post-dose
Pharmacokinetics: Pharmacokinetic lag time (Tlag) | Up to 60 hours post-dose
  Tlag is defined as the time of observation prior to the first observation with a measurable (non-zero) concentration.
Pharmacokinetics: Time of maximum observed plasma concentration (Tmax) | Up to 60 hours post-dose
Pharmacokinetics: Area under the plasma concentration-time curve from time zero up to time t (AUCt) | Up to 60 hours post-dose
  AUCt is defined as the area under the plasma concentration-time curve from time zero up to time t, where t is the last time point at which the concentration is above the lower limit of quantification (time of last measurable [non-zero] concentration [tlast]).
Pharmacokinetics: Area under the plasma concentration-time curve to infinity (AUCinf) | Up to 60 hours post-dose
Pharmacokinetics: %Extrap AUC | Up to 60 hours post-dose
  %Extrap AUC is defined as the percentage of AUC that is due to extrapolation from the last measurable concentration.
Pharmacokinetics: Terminal half-life (t1/2) | Up to 60 hours post-dose
Pharmacokinetics: Terminal elimination rate constant (λz) | Up to 60 hours post-dose
  λz is defined as the first-order rate constant associated with terminal (log-linear) portion of the plasma concentration-time curve estimated via linear regression of the time versus log concentration.
Pharmacokinetics: Apparent total systemic clearance (CL/F) | Up to 60 hours post-dose
Pharmacokinetics: Apparent volume of distribution associated with the terminal phase (VZ/F) | Up to 60 hours post-dose
Pharmacokinetics: Mean residence time (MRT) | Up to 60 hours post-dose
Number of subjects with adverse events (AEs) and type of adverse events | From screening (Day-28 to Day -1) up to the end-of-study (Day 3)
  An AE is defined as any untoward medical occurrence in a subject taking part in a clinical study. Number of subjects with any AE (serious or non-serious) are presented.
Number of subjects with abnormal laboratory parameters | From screening (Day-28 to Day -1) up to the end-of-study (Day 3)
  Number of subjects with abnormal findings in laboratory parameters (biochemistry, hematology, and urine analysis) will be presented.
Number of subjects with abnormal vital signs | From screening (Day-28 to Day -1) up to the end-of-study (Day 3)
  Number of subjects with abnormal findings in vital signs will be presented.
Number of subjects with abnormal changes in ECG | From screening (Day-28 to Day -1) up to the end-of-study (Day 3)
  Number of subjects with abnormal findings in ECG will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India